CLINICAL TRIAL: NCT04815343
Title: Investigation of the Naída CI M90 Sound Processor in Various Acoustic Scenarios
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Bionics AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ABIntl-20-04
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: comparision of different conditions with-in subject. (10 bimodal, 10 bilateral CI users)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral users (Experimental): two implant systemswith two sound processors
  Interventions: Device: Naída CI M90 Sound Processor (hearing aid and cochlea implant sound processor)
- Bimodal user (Experimental): with one sound processor and one hearing aid
  Interventions: Device: Naída CI M90 Sound Processor (hearing aid and cochlea implant sound processor)

INTERVENTIONS:
Device: Naída CI M90 Sound Processor (hearing aid and cochlea implant sound processor) — Speech perception measures, Hearing thresholds, Enjoyment rating, Sound identification, Subjective feedback

SUMMARY:
In this clinical trial, an un-controlled, repeated measures open design with within-subject comparison will be used to evaluate the effect of Naída Link M90 hearing aid and Naída CI M90 sound processor on sound perception. This design was shown to be successful in previous studies for the evaluation of sound coding strategies. Furthermore, a within-subject comparison decreases the variance in the results allowing for fewer subjects when the population that uses the investigational device is not large in general.

ELIGIBILITY:
Inclusion Criteria:

* CI users with a CII, HiRes90K (Advantage) or HiRes Ultra implant system

  * Bilateral users: two implant systems
  * Bimodal users: hearing aid contralateral
* Minimum of 18 years of age
* Minimum of six months experience with their implant system
* Minimum of six months experience with the Naída CI Q-Series sound processor
* Ability to give feedback on sound quality
* Speech intelligibility with the HSM sentence test in noise at 10 dB SNR > 10% as obtained during previous visits in the clinical routine
* Fluent in German language

Exclusion Criteria:

* Difficulties additional to hearing impairment that would interfere with the study procedures
* Concurrent participation in other study
* Pregnant and breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Difference in speech perception in noise with AutoSense OS on Naída M hearing devices and AutoSound OS on the clinically available Naída Q hearing devices | 6 weeks
  Difference in speech reception threshold of 50% speech understanding which is the signal to noise ratio in Decibel [dB] to understand 50% of the target speech between AutoSense OS on Naída M hearing devices and AutoSound OS on the clinically available Naída Q hearing devices.

SECONDARY OUTCOMES:
Differences in speech perception in noise threshold measured in Decibel [dB] | 6 weeks
  Differences are compared between AutoSense OS on Naída M hearing devices and the omnidirectional microphone setting on Naída Q hearing devices.
  Min and Max values are -10dB and +10dB, whereas the smalller the value the better
Differences in speech perception in quiet threshold measured in Decibel [dB] | 6 weeks
  Differences are compared between AutoSense OS on Naída M hearing devices and AutoSound OS on Naída Q hearing devices and the omnidirectional microphone setting on Naída Q hearing devices.
  Min and Max values are -10dB and +10dB, whereas the smalller the value the better
Differences in mono/stereo identification measured in % correct | 6 weeks
  Differences are compared between mono and stereo free-field presentation, mono and stereo streaming presentation, stereo free-field and stereo streaming presentation, mono free-field and mono streaming presentation, differences in music enjoyment ratings measured in rating score
Differences in speech understanding in noise measured in % correct | 6 weeks
  Differences are compared between AutoZoomControl on Naída M hearing devices and the omnidirectional microphone setting on Naída Q hearing devices
Differences in music enjoyment ratings measured in rating score | 6 weeks
  Differences are compared between
  * mono and stereo free-field presentation
  * mono and stereo streaming presentation
  * stereo free-field and stereo streaming presentation
  * mono free-field and mono streaming presentation

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No